CLINICAL TRIAL: NCT05558423
Title: The Intermittent Fasting ZOE Health Study: Effects on Hunger, Mood, Energy and Symptom Burden in a UK Cohort
Brief Title: ZOE Health Study: The Intermittent Fasting Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zoe Global Limited (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZHS-IF
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-09

CONDITIONS: Intermittent Fasting; Time Restricted Feeding
Keywords: Intermittent Fasting; Time Restricted Eating; Hunger; Mood; Energy
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-controlled (Experimental): n-of-1 design. Participants complete a baseline habitual eating phase following by an intervention TRE phase.
  Interventions: Behavioral: Time Restricted Eating

INTERVENTIONS:
Behavioral: Time Restricted Eating — Participants are asked to follow a Time Restricted Eating regimen with eating window of ≤10 hours.

SUMMARY:
The timing of food intake (chrononutrition) is emerging as a key regulator of circadian rhythm in metabolic organs. A wealth of research has been conducted on intermittent fasting, and time restricted eating (TRE) specifically, investigating the temporal patterns of diet (eating window, time of eating, time of largest energy intake) and their impact on disease risk, with overall beneficial impact on health. Studies have been conducted in a parallel or single arm design, while cross-over and the efficacy of TRE in ameliorating appetite and symptom burden within an individual remains unclear.

DETAILED DESCRIPTION:
Time Restricted Eating (TRE; a type of intermittent fasting) is a dietary pattern based on the 24h day. Practicing individuals restrict their eating/feeding window to a certain number of hours, e.g. 4h, while the remaining hours in the day are non-feeding (fasting) time. The eating window is the duration of time from the start of the first meal to the end of the last meal in a 24 hr period. The eating window in a general population has previously been quantified at 12h (American cohort of n=15,000). It is important to note that TRE differs from other intermittent fasting protocols by (i) not specifying a change in dietary intake, such as requiring caloric restriction, but rather specifying the temporal pattern of intake; and (ii) requiring consistent daily eating windows over several days. TRE protocols can vary in the length of the eating window, as well as the anchoring of that window to the time of day, such that early vs. middle vs. late TRE regimens exist.

While the cardiometabolic benefits TRE are well established by human trials, other outcomes of dietary compliance remain unexplored and thus bring into question the sustainability of and adherence to TRE as a long-term dietary regimen. Perception of hunger, mood and energy, and self-elected timings of TRE eating windows while following the dietary pattern are not well understood. In particular, the relative differences in these outcomes between an habitual and a TRE eating pattern within the same individual must be determined in order to truly evaluate the acceptability of TRE on a per-individual basis.

The Intermittent Fasting Study, a sub-study of the ZOE Health Study (ZHS), will test the effects of habitual eating patterns vs. a TRE protocol on hunger, mood, energy and symptom burden in an adult UK cohort using the ZHS app.

Population:

This study is open to all participants currently enrolled in the ZHS study tracking physical and mental symptom burden on a daily basis. Participants will be invited to take part in the Intermittent Fasting Study and must provide their consent in order to participate.

Design:

The study will take place remotely using a n-of-1 design, consisting of two phases with a non-randomised cross-over. Firstly, the participant will complete a baseline phase of one week, where they follow their habitual eating pattern.

Secondly, for the second and third weeks of the study, the participant will be asked to follow a TRE regimen with an eating window of ≤10 hours. The exact duration of the eating window, its timing relative to time of day, and participant dietary intake, are decisions deliberately left to the participant for two reasons; (i) to enable the participant to choose exactly the right TRE protocol that is most acceptable to them and therefore most likely to be sustainable in the long-term; (ii) to understand the trends in acceptability and feasibility of TRE regimens across this UK cohort. The participant is given the option of continuing their TRE phase beyond the minimum two weeks.

During the two phases, participants are asked to log the following outcomes in the ZHS app, on a daily basis:

* Hunger (using visual analogue scales, VAS)
* Mood (using VAS)
* Energy (using VAS)
* Symptom burden (using VAS)
* Body weight (optional)
* Clock time of the start of their first eating event
* Clock time of the end of their last eating event

Participants may also be asked to log their diet during their baseline phase and their TRE phase (optional) such that the temporal effect of changing between their habitual and chosen TRE regimens on dietary intake can be determined. They will also be asked to complete questionnaires, at the start and end of the study, about their eating habits, gastrointestinal health, lifestyle and demographic.

Outcome analysis may be stratified according to demographic and other exposure parameters such as early vs. late TRE.

ELIGIBILITY:
Participants on the ZOE Health Study (ZHS) app are accepted onto the study if they wish to participate and are within the UK.

The ZHS eligibility criteria are as follows:

Inclusion Criteria:

* Adults of 18 years and above, where the app has been approved for download from the Apple App and Google Play stores.

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150000 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2023-10-24 (Estimated)

PRIMARY OUTCOMES:
TRE window clock time | 2 weeks
  The chosen clock time for the TRE window (early, vs. middle, vs. late)
Habitual eating window clock time | 1 weeks
  The chosen clock time for the habitual eating window
Hunger | 3 weeks (plus optional unlimited weeks)
  Hunger levels reported by visual analogue scale ("how hungry did you feel yesterday?"; 0-10; where 10 is the most hungry)
Mood | 3 weeks (plus optional unlimited weeks)
  Mood levels reported by visual analogue scale ("how was your mood yesterday?"; 0-10; where 10 is most positive)
Energy | 3 weeks (plus optional unlimited weeks)
  Energy levels reported by visual analogue scale ("how energetic did you feel yesterday?"; 0-10; where 10 is most energetic)
Symptom burden | 3 weeks (plus optional unlimited weeks)
  The self-reported symptom burden while completing both habitual and TRE phases

SECONDARY OUTCOMES:
Body weight | 3 weeks (plus optional unlimited weeks)
  Self-reported in the study app (optional)
Gastrointestinal symptoms | 3 weeks (plus optional unlimited weeks)
  Gastrointestinal symptoms self-reported by questionnaire
Eating habits | 3 weeks (plus optional unlimited weeks)
  Eating habits self-reported by questionnaire, including number of main meals and snacks per day

CONTACTS AND LOCATIONS:
Overall Officials: Tim Spector, Pr, Principal Investigator — Zoe Ltd, King's College London
Locations (1):
- ZOE Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No